CLINICAL TRIAL: NCT02740582
Title: Effects of Tolcapone on Decision Making and Alcohol Intake Using a Laboratory Bar in Moderate to Heavy Social Drinkers
Brief Title: Effects of Tolcapone on Decision Making and Alcohol Intake in Alcohol Users
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Mitchell (Other)
Responsible Party: Sponsor-Investigator, Jennifer Mitchell, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Tolcapone Lab Bar
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Alcohol Abuse; Impulsive Behavior
MeSH Terms: conditions — Alcoholism; Impulsive Behavior | interventions — Tolcapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tolcapone First, then Placebo (Experimental): Tolcapone arm first: 5 days of 100 mg tolcapone TID, followed by washout period, then 5 days of placebo TID
  Interventions: Drug: Tolcapone; Drug: Placebo
- Placebo First, then Tolcapone (Placebo Comparator): Placebo arm first: 5 days placebo, followed by washout period, followed by 5 days of 100 mg tolcapone TID
  Interventions: Drug: Tolcapone; Drug: Placebo

INTERVENTIONS:
Drug: Tolcapone
  Other Names: Tasmar
Drug: Placebo

SUMMARY:
The purpose of this study is to determine the effects of tolcapone on decision making and alcohol intake using a laboratory bar (on-site alcohol self-administration) in alcohol drinkers.

DETAILED DESCRIPTION:
The study is a 7-session, double blind, placebo-controlled crossover study of the effects of tolcapone, the COMT inhibitor, on decision making and alcohol intake using a laboratory bar in moderate to heavy social alcohol drinkers. Subjects will be moderate to heavy social users of alcohol, defined as at least 10 standard drinks per week for women and at least 14 standard drinks per week for men. There will be one screening session followed by six additional visits including 2 laboratory bar sessions. On each study drug administration day, subjects will come in to the clinic for a medication dispensation visit and instructions on when and how to take the study drug for the remainder of the study. Study drug bottles will be equipped with MEMS caps to ensure compliance. After 5 days of drug administration, subjects will return to the clinic for a laboratory bar. This session will consist of administration of a standardized laboratory bar paradigm and a series of computerized and written decision-making tasks. Subjects will then be crossed over and complete the same series of study visits on the alternate study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who are 21-40 years of age
* If female, 10 or more alcoholic drinks must be consumed weekly.
* If male, 14 or more alcoholic drinks must be consumed weekly.
* Meets DSM-V criteria for Alcohol Use Disorder (AUD).
* If female, must be non-lactating, not pregnant, and using a reliable contraception method (i.e. abstinence, intrauterine device [IUD], hormonal birth control, or barrier method).
* Ability to read and speak English.
* High school graduate.
* Able and willing to provide an informed consent.
* Able to understand and follow the instructions of the investigator, including the delayed discounting tasks. Residing within 5 miles of the study site.

Exclusion Criteria:

* Positive urine drug screen (except marijuana).
* Using cocaine, stimulants (other than nicotine and caffeine), amphetamines, hallucinogens, ecstasy, opiates, sedatives, pain pills, sleeping pills. or other psychoactive drugs within 2 weeks of the start of the study (except marijuana).
* Marijuana use more than 3 times/week.
* Current enrollment in an alcohol, or other drug treatment program or current legal problems relating to alcohol, or other drug use.
* Currently trying to quit alcohol use.
* History of major alcohol related complications within the preceding 2 years (liver failure/cirrhosis, pancreatitis, esophageal varices, etc.).
* Two SGPT/ALT or SGOT/AST values greater than the upper limit of normal.
* Unable to pass the Standard Field Sobriety Test in a sober state (BAC = 0.00).
* BAC level >0.05% at the beginning of screening visit (within margin of error of detection).
* Regular use of any of the drugs on the tolcapone contraindications list OR within 2 weeks of drug administration.
* Severe low blood (< 90/50) pressure or uncontrolled high blood pressure (>160/100). Allergy or intolerance to tolcapone.
* Subject has received an investigational drug within 30 days of the screening visit.
* Subject is considered unsuitable for the study in the opinion of the investigator or clinician for any other reason (such as an Axis II personality disorder that makes the subject unable to comply with study instructions, per the Clinician's judgement.)

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mitchell, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, Berkeley, Berkeley, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Result] Coker AR, Weinstein DN, Vega TA, Miller CS, Kayser AS, Mitchell JM. The catechol-O-methyltransferase inhibitor tolcapone modulates alcohol consumption and impulsive choice in alcohol use disorder. Psychopharmacology (Berl). 2020 Oct;237(10):3139-3148. doi: 10.1007/s00213-020-05599-5. Epub 2020 Jul 2. PMID 32617646

RESULTS

PARTICIPANT FLOW:
Groups:
- Tolcapone First: Tolcapone arm first: 5 days of 100 mg tolcapone TID, followed by washout period, then 5 days of placebo TID
- Placebo First: Placebo arm first: 5 days placebo, followed by washout period, followed by 5 days of 100 mg tolcapone TID
Period: First Intervention
Arm/Group | Tolcapone First | Placebo First
Started | 29 | 33
Completed | 24 | 31
Not Completed | 5 | 2
Period: Washout
Arm/Group | Tolcapone First | Placebo First
Started | 24 | 31
Completed | 24 | 31
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Tolcapone First | Placebo First
Started | 24 | 31
Completed | 23 | 28
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Population: Completers of study were used for analysis
Groups:
- Tolcapone First: Tolcapone arm first: 5 days of 100 mg tolcapone TID, followed by washout period, then 5 days of placebo TID
  Tolcapone
  Placebo
- Placebo First: Placebo arm first: 5 days placebo, followed by washout period, followed by 5 days of 100 mg tolcapone TID
  Tolcapone
  Placebo
- Total: Total of all reporting groups
Arm/Group | Tolcapone First | Placebo First | Total
Number analyzed (Participants) | 23 | 28 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 28 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 24.4 [21 to 32] | 27.3 [21 to 35] | 25.98 [21 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 14 | 22
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 20 | 23 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 15 | 18 | 33
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 28 | 51
Self-reported alcoholic drinks / week [Mean (Full Range); unit: alcoholic drinks / week] | 24.79 [10 to 52] | 18.13 [10 to 49.5] | 21.13 [10 to 52]

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinks Consumed in a Laboratory Bar Session
Description: Number of drinks consumed in a laboratory bar session (out of a maximum of 4 drinks available) following either placebo or tolcapone administration.
Time Frame: A laboratory bar session is 1 hour long
Population: Completers were analyzed
Measure: Mean (Standard Deviation); unit: drinks
Groups:
- Tolcapone First, Then Placebo: Tolcapone arm first: 5 days of 100 mg tolcapone TID, followed by washout period, then 5 days of placebo TID
  Tolcapone
  Placebo
- Placebo First, Then Tolcapone: Placebo arm first: 5 days placebo, followed by washout period, followed by 5 days of 100 mg tolcapone TID
  Tolcapone
  Placebo
Arm/Group | Tolcapone First, Then Placebo | Placebo First, Then Tolcapone
Number analyzed (Participants) | 23 | 28
drinks
  Drinks on Placebo | 2.69 (1.45) | 2.96 (1.1)
  Drinks on tolcapone | 2.73 (1.38) | 2.39 (1.66)

ADVERSE EVENTS:
Time Frame: From enrollment through study completion, an average of 3 weeks
Description: The study staff will probe, via effects scale survey completed by subjects and discussion with the subject where necessary, for the occurrence of AEs during each subject visit. Study staff will continue to follow up with the subject daily until the matter is resolved (AE has decreased to 2).
Groups:
- Tolcapone: Adverse Events Groups are being reported "per intervention" (e.g., "Tolcapone" and "Placebo") rather than based on group in the cross over study. Tolcapone Group here reflect all participants who received Tolcapone during the study, regardless of order.
- Placebeo: Adverse Events Groups are being reported "per intervention" (e.g., "Tolcapone" and "Placebo") rather than based on group in the cross over study. Placebo Group here reflect all participants who received Placebo during the study, regardless of order.
Arm/Group | Tolcapone | Placebeo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/57
Other Adverse Events (participants affected / at risk) | 0/60 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT02740582/Prot_SAP_000.pdf